CLINICAL TRIAL: NCT02009410
Title: A Double-blind, Randomized, Multi-center, Placebo-controlled, Parallel-group Study to Assess the Effect of Creon® on Pancreatic Exocrine Insufficiency in Subjects With Diabetes Mellitus Type 2
Brief Title: A Study to Assess the Effect of Creon® on Pancreatic Exocrine Insufficiency in Subjects With Diabetes Mellitus Type 2
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Nuvisan (Unknown); Datamap (Industry); ClinIntel (Industry); Catalent (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-954; 2013-001347-31 (EudraCT Number)
Record Dates: First submitted 2013-11-25; First posted 2013-12-12 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Exocrine Pancreatic Insufficiency in Subjects With Diabetes Mellitus Type 2
Keywords: Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Creon (Experimental)
  Interventions: Drug: Creon
- Placebo (Placebo Comparator)
  Interventions: Drug: Creon 25000 matching Placebo

INTERVENTIONS:
Drug: Creon — Creon 25000 (2 capsules per meal 3 times per day and 1 capsule/snack 2 times per day) during 12 weeks
  Arms: Creon
Drug: Creon 25000 matching Placebo — Creon 25000 placebo matching capsules (2 capsules per meal 3 times per day and 1 capsule/snack 2 times per day) during 12 weeks
  Arms: Placebo

SUMMARY:
maldigestion of dietary macronutrients (pancreas not producing enough enzymes for digestion of fat, sugars and proteins) in diabetes type II

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* BMI < 30 kg/m2
* History of type 2 diabetes mellitus as confirmed by:
* onset of diabetes after 30 years of age and
* no insulin treatment in the first year after diagnosis
* Subjects on insulin treatment or on insulin treatment in combination with oral antidiabetics
* HbA1c > 6.5% in medical history within the last 6 months despite insulin treatment
* Not previously treated with any pancreatic enzyme supplementation

Inclusion Criterion at Visit 1:

• FE-1 (fecal elastase 1) <100μg/g of stool

Inclusion Criterion at Visit 2:

• 13C MTBT of <29% 13CO2-CRR (Carbon dioxide-Cumulative Recovery Rate)

Exclusion Criteria:

* Treatment with systemic steroids for at least 3 weeks within past 6 months
* Patients with a known pancreatic exocrine insufficiency due to non-diabetic diseases, e.g., chronic pancreatitis, pancreatectomy, cystic fibrosis, celiac disease, shwachman-diamond syndrome, gastrectomy, etc.
* Any type of malignancy involving digestive tract in the last 5 years
* Any type of gastrointestinal surgery (except appendectomy and gallbladder resection)
* Short bowel syndrome
* Hemochromatosis
* Known late onset autoimmune diabetes in the adult
* Any history of drug abuse including alcohol
* Positive urine pregnancy test; lactation; females of child-bearing potential who are not using either an oral hormonal contraceptive or an intrauterine device
* Hypersensitivity to the active substance or to any of the excipients
* Intake of an experimental drug within 4 weeks prior to entry into this study
* Suspected non-compliance or non-cooperation
* History of human immunodeficiency virus (HIV) infection

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Recovery rate of 13CO2 (carbon dioxide with stable isotope of carbon) | from baseline up to the week 12 visit

SECONDARY OUTCOMES:
Change in nutritional parameters | from baseline up to the week 12 visit
  fat soluble vitamins (D and E), retinol-binding protein, albumin, pre-albumin, magesium and calcium will be measured.
Change in HbA1c | from baseline up to the week 12 visit
Change in quality of life assessed via a questionnaire Gastrointestinal-Quality of Life Index (GIQL) | from baseline up to the week 12 visit
Change in clinical global impression of disease symptoms | from baseline up to the week 12 visit
  disease symptoms will be rated by the subject according a rating scale

OTHER OUTCOMES:
vital signs | from baseline up to the week 12 visit
  blood pressure and heart rate, body weight and BMI
routine safety laboratory | from baseline up to the week 12 visit
  Hematology, biochemistry and a urine pregnancy test will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Suntje Sander-Struckmeier, PhD, Study Director — Abbott
Locations (10):
- Germany (4):
  - Site reference no. 113456, Bochum
  - Site reference no. 113477, Frankfurt
  - Site reference no. 113476, Pohlheim
  - Site reference no. 113475, Ulm
- Spain (6):
  - Site reference no. 112517, Ávila
  - Site reference no. 112519, Madrid
  - Site reference no. 112520, Málaga
  - Site reference no. 112495, Santiago de Compostela
  - Site reference no. 112518, Segovia
  - Site reference no. 112496, Seville